CLINICAL TRIAL: NCT07248254
Title: Effects of Wilbarger Deep Pressure and Proprioceptive Technique (DPPT) on Motor Skills and Sleep Pattern in Children With Autism Spectrum Disorder.
Brief Title: Effects Of DPPT On Motor Skills And Sleep In Children With Autism
Acronym: DPPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REC/RCR&AHS/AIZAZAMIR
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Wilbarger Protocol, DPPT, Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: A quasi-experimental study will be conducted across pediatric therapy centers, autism clinics, and special schools using convenience sampling. Autistic children aged 6-10 years with sensory processing difficulties, motor delays, and sleep disturbances will be included, excluding those with other neurological or major physical disorders. Motor skills will be assessed using the BOT-2 and sleep quality with the CSHQ. Participants will receive the Wilbarger DPPT along with routine therapies (e.g., OT, PT, ABA) three times weekly for six weeks (30-45 min/session). Data will be collected at baseline and post-intervention to assess motor and sleep improvements. Statistical analysis will be performed using SPSS v23.
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Other): Participants will receive the Wilbarger Deep Pressure and Proprioceptive Technique (DPPT) along with their usual therapies (OT, PT, ABA) to improve sensory processing, motor skills, and sleep in children with ASD. Sessions will be conducted in a calm setting, with explanations provided to ensure comfort. The DPPT includes 5-10 minutes of deep-pressure brushing using a soft surgical brush on the arms, back, legs, and feet, followed by 5-10 minutes of gentle joint compressions on shoulders, elbows, knees, and ankles (3-5 seconds each). Calming activities like deep breathing or quiet play will follow to aid sensory integration. The intervention will occur thrice weekly for six weeks (30-45 minutes/session). Progress will be measured using BOT-2 for motor skills and CSHQ for sleep at baseline and post-intervention.
  Interventions: Other: Wilbarger Deep Pressure and Proprioceptive Technique (DPPT)

INTERVENTIONS:
Other: Wilbarger Deep Pressure and Proprioceptive Technique (DPPT) — Participants will receive the Wilbarger Deep Pressure and Proprioceptive Technique (DPPT). Each session will begin in a calm, quiet environment to reduce distractions, with the therapist explaining the process in simple terms. The brushing protocol involves using a soft surgical brush to apply firm yet gentle deep pressure to the arms, back, legs, and feet for about 5-10 minutes. This is followed by gentle joint compressions to the shoulders, elbows, knees, and ankles, each held for 3-5 seconds, lasting another 5-10 minutes. Afterward, calming activities such as deep breathing or quiet play help the child integrate the sensory input. The DPPT will be administered three times per week for six weeks, with each session lasting approximately 30-45 minutes, including brushing, joint compressions, and calming activities.

SUMMARY:
It will be conducted as a Quasi Experimental study across pediatric therapy centers, specialized autism clinics, and special schools. Using non-probability convenience sampling, the study will enroll Autistic children aged 6-10 years who exhibit sensory processing difficulties, motor skill delays, and sleep disturbances. Exclusion criteria include other neurological or developmental disorders and children with major physical problems. Motor skills will be assessed with the Bruininks-Oseretsky Test of Motor Proficiency (BOT-2), and sleep quality will be measured using the Children's Sleep Habits Questionnaire (CSHQ).

Participants will be receiving Wilbarger DPPT along with their usual therapy sessions, which may include general occupational therapy, physical therapy, ABA etc. The DPPT intervention will occur three times per week for six weeks, with each session lasting approximately 30-45 minutes, including brushing, joint compressions, and calming activities. Data will be collected at baseline and post-intervention, focusing on motor skill improvement and sleep quality changes. SPSS version 23 will be used for statistical analysis.

DETAILED DESCRIPTION:
Children with Autism Spectrum Disorder (ASD) frequently experience sensory processing difficulties, where they may either overreact or underreact to sensory stimuli in their environment. This sensory deregulation can significantly impact essential functions, including motor skills and sleep quality, both0 crucial for overall development and day-to day engagement. Sensory Integration Therapy (SIT), is a well-established approach used to help individuals with sensory processing challenges. Ayres' work emphasized that when the brain effectively organizes sensory input, it can foster better behavioral and motor responses, leading to improved participation in daily activities. Various sensory-based interventions have been developed, including Wilbarger Deep Pressure and Proprioceptive Technique (DPPT). The Wilbarger protocol, or DPPT, is a specific approach using firm pressure and joint compressions at regular intervals, aiming to create a calming, organizing effect on the nervous system. The "brushing" aspect of this technique involves using a soft surgical brush over the skin to stimulate sensory receptors, followed by compressions to the joints, which is thought to help regulate sensory input and reduce sensory defensiveness. This study aims to assess the impact of DPPT on motor skills and sleep patterns in children with ASD, exploring whether DPPT can enhance functional motor skills and improve sleep quality.

It will be conducted as a Quasi Experimental study across pediatric therapy centers, specialized autism clinics, and special schools. Using non-probability convenience sampling, the study will enroll Autistic children aged 6-10 years who exhibit sensory processing difficulties, motor skill delays, and sleep disturbances. Exclusion criteria include other neurological or developmental disorders and children with major physical problems. Motor skills will be assessed with the Bruininks-Oseretsky Test of Motor Proficiency (BOT-2), and sleep quality will be measured using the Children's Sleep Habits Questionnaire (CSHQ).

Participants will be receiving Wilbarger DPPT along with their usual therapy sessions, which may include general occupational therapy, physical therapy, ABA etc. The DPPT intervention will occur three times per week for six weeks, with each session lasting approximately 30-45 minutes, including brushing, joint compressions, and calming activities. Data will be collected at baseline and post-intervention, focusing on motor skill improvement and sleep quality changes. SPSS version 23 will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with Autism
* Both Genders Males and Females
* Age 6-11
* Autistic children diagnosed with sensory processing disorder and reported with motor skill delays and sleep disturbances.
* Children scoring within the "Definite Difference" range in sensory processing areas on the Sensory Profile 2.

Exclusion Criteria:

* Children with other neurological or Developmental disorders
* No serious physical or behavioral impairments (blindness and deafness)
* Children with multiple diagnosis along with ASD.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Bruininks-Oseretsky test for Motor Proficiency (BOT-2) | Baseline,6 weeks
  The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) is an individually administered test that uses engaging, goal-directed activities to measure a wide array of motor skills in individuals ages 4 through 21. The BOT-2 uses a subtest and composite structure that highlights motor performance in the broad functional areas of stability, mobility, strength, coordination, and object manipulation.
Children Sleep Habits Questionnaire (CSHQ) | Baseline,6 weeks
  The Children's Sleep Habits Questionnaire (CSHQ) is one of the most commonly used assessment tools for pediatric sleep. It is used both in research and in the clinical field. The CSHQ is a 45-item questionnaire. Each question on the questionnaire is rated on a 3-point scale based on the frequency of occurrence within the past week.
  Resp Sets are categorized as ''usually'' (5-7 times within the past week), ''sometimes'' (2-4 times within the past week), or ''rarely (never of 1 time within the past week). Some items on the questionnaire are reverse-scored, ensuring that higher scores consistently indicate problem behaviors. All responses are totaled to create a Total Sleep Disturbance index (range from 33 99), with a score exceeding 41 suggesting the presence of a pediatric sleep disorder.

CONTACTS AND LOCATIONS:
Overall Officials: AIZA ZAMIR, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Mind Care Therapy Centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoen SA, Schaaf RC, Mailloux Z, Bundy A, Lane S, May-Benson TA, Parham LD, Roley SS. Response: Commentary: Evaluating Sensory Integration/Sensory Processing Treatment: Issues and Analysis. Front Integr Neurosci. 2022 Jun 7;16:874320. doi: 10.3389/fnint.2022.874320. eCollection 2022. No abstract available. PMID 35747497